CLINICAL TRIAL: NCT06987279
Title: Lactobacillus Plantarum Lp90 and Hormonal Regulation in Obese Women：A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Lactobacillus Plantarum and Hormonal Regulation in Obese Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WK20250515
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Women
MeSH Terms: conditions — Obesity | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Take Lactobacillus plantarum Lp90 at 30 billion CFU per day.
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Taking maltodextrin 3 g/day.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial period of this study is 3 months, and each patient will undergo 4 visits (in month 0, month 1, month 2, and month 3).
  Arms: Probiotic Group
Dietary Supplement: Maltodextrin — The trial period of this study is 3 months, and each patient will undergo 4 visits (in month 0, month 1, month 2, and month 3).
  Arms: Placebo Group

SUMMARY:
To evaluate the regulatory effect of Lactobacillus plantans Lp90 formula on visceral fat metabolism and sex hormone balance in obese women.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 40 years old, female, BMI ≥ 25 kg/m2.
2. Be willing to receive follow-up during the intervention period.
3. Be willing to provide two blood, urine and fecal samples during the intervention period.
4. Be willing to take the compound probiotics by oneself every day during the intervention period.
5. Have good hearing and be able to hear and understand all instructions during the intervention period.

   -

Exclusion Criteria:

1. Suffering from digestive system diseases, mainly gastrointestinal diseases (celiac disease, ulcerative colitis, Crohn's disease).
2. Suffering from severe neurological disorders (epilepsy, stroke, severe head trauma, meningitis within the past 10 years, brain surgery, brain tumor, long-term coma - excluding general anesthesia).
3. Have received/are currently receiving treatment for the following mental illnesses: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder.
4. Take medication for depression or low mood.
5. Suffering from internal organ failure (such as heart, liver or kidney failure, etc.).
6. Have received radiotherapy or chemotherapy in the past.
7. Have received general anesthesia surgery/procedures within the past three years, or plan to receive general anesthesia procedures/surgeries within the next three months during this trial.
8. Have suffered from hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past.

   -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The changes of estradiol before and after the intervention | 0, 1, 2, 3 months
  The serum estrogen content of the subjects before and after the intervention was detected by enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Central-China Cardiovascular Hospital, Zhengzhou, Henan, China